CLINICAL TRIAL: NCT05815836
Title: Precision Medicine in Stroke
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Steffen Tiedt, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: LMU_ISD_2023_PROMISE
Record Dates: First submitted 2023-03-09; First posted 2023-04-18 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Brain Ischemia; Nervous System Diseases
Keywords: Biomarker; Stroke; Diagnosis; Pathophysiology
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Brain Ischemia; Nervous System Diseases; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, platelet-poor plasma, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute Ischemic Stroke: 504 patients admitted to a specialized stroke service because of an acute ischemic stroke. The circulating proteome and metabolome as well as specific molecular targets of interest (i.e. NfL) will be assessed upon admission (day 1), the next morning (day 2), day 3, day 7 (or day of discharge if earlier), and day 90. Routinely collected clinical data including from neuroimaging will be collected throughout hospitalization. Clinical follow-up will be performed at 3 months.
- Acute Intracerebral hemorrhage: 130 patients admitted to a specialized stroke service because of an acute intracerebral hemorrhage. The circulating proteome and metabolome as well as specific molecular targets of interest (i.e. NfL) will be assessed upon admission (day 1). Routinely collected clinical data including from neuroimaging will be collected throughout hospitalization.
- Stroke Mimics: 51 patients admitted to the emergency department because of acute stroke-like symptoms caused by epileptic seizures, migraine attacks, or other stroke-mimicking diseases. The circulating proteome and metabolome as well as specific molecular targets of interest (i.e. NfL) will be assessed upon admission (day 1), the next morning (day 2), day 3, day 7, and day 90. Routinely collected clinical data including from neuroimaging will be collected throughout hospitalization.
- Healthy subjects: 102 subjects without acute neurological symptoms. The circulating proteome and metabolome as well as specific molecular targets of interest (i.e. NfL) will be assessed.

SUMMARY:
PROMISE aims at identifying novel diagnostic and prognostic circulating biomarkers for patients with acute stroke and at informing on crucial yet undetected pathophysiological mechanisms driving outcome after stroke by enriching all phenotypic information available from clinical routine with in-depth quantification of the circulating proteome and metabolome as well as other entities.

DETAILED DESCRIPTION:
The heterogeneity of ischemic stroke (IS) poses a challenge for assigning patients to optimal treatment strategies and is a major reason for the large number of failed clinical trials. Current diagnostic algorithms are insufficient to explain clinical outcomes arguing for crucial yet undetected pathophysiological mechanisms. Diagnostic tests further leave stroke etiology undetermined in 40 % of IS patients thus impeding the allocation of these patients to optimal secondary prevention regimens. Heterogeneity is also seen at the level of neuronal injury, which greatly varies between IS patients, but can neither be assessed in the pre-hospital setting nor serially in the acute phase to monitor stroke progression and to develop individual trajectories of neuronal loss over time. The circulating proteome and metabolome capture pathophysiological events from multiple organs including local and systemic events (e.g. stress) related to acute stroke and might thus inform on neuronal injury and the mechanisms causing stroke. The circulating proteome and metabolome may further inform on i) the systemic effects of stroke, which contribute significantly to stroke outcome but are under-researched, and ii) how concepts from preclinical stroke research such as reperfusion injury translate to human stroke. The investigators hypothesize that the combination of detailed clinical phenotyping with advanced profiling technologies (genomics, proteomics, and metabolomics) will enable the identification of key molecular signatures of IS that inform on pathophysiological mechanisms and might also be utilized as diagnostic instruments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke:
* Age 18 years or older
* Diagnosis of an acute ischemic stroke defined by an acute focal neurological deficit in combination with a diffusion-weighted imaging-positive lesion on magnetic resonance imaging or a new lesion on a delayed CT scan.
* Time from last seen well to admission and first blood sampling < 24 hours
* Blood samples collected upon admission (day 1), the next morning (day 2), day 3, and day 7 (or day of discharge if earlier)
* Informed consent in accord with ethical approval
* Patients with acute intracerebral hemorrhage:
* Age 18 years or older
* Diagnosis of an acute intracerebral hemorrhage defined by an acute focal neurological deficit in combination with imaging-based evidence of intracerebral hemorrhage.
* Time from last seen well to admission and first blood sampling < 24 hours
* Blood samples collected upon admission (day 1)
* Informed consent in accord with ethical approval
* Patients with stroke mimics:
* Age 18 years or older
* Diagnosis of a stroke-mimicking disease defined by an acute focal neurological deficit in combination with a lack of infarction on neuroimaging.
* Time from last seen well to admission and first blood sampling < 24 hours
* Blood samples collected upon admission (day 1), the next morning (day 2), day 3, and day 7
* Informed consent in accord with ethical approval
* Healthy subjects:
* Age 18 years or older
* Informed consent in accord with ethical approval

Exclusion Criteria:

* Patients with acute ischemic stroke:
* Lack of follow-up CT or MRI imaging
* Major surgery within the last four weeks
* In-house stroke
* Myocardial infarction, ischemic stroke, transient ischemic attacks, traumatic brain injury, cerebral venous sinus thrombosis, any intracranial hemorrhage, thrombosis, or pulmonary embolism within the last four weeks
* Chronic inflammatory bowel disease or percutaneous endoscopic gastrostomy
* Patients with acute intracerebral hemorrhage:
* Major surgery within the last four weeks
* In-house stroke
* Myocardial infarction, ischemic stroke, transient ischemic attacks, traumatic brain injury, cerebral venous sinus thrombosis, any intracranial hemorrhage, thrombosis, or pulmonary embolism within the last four weeks
* Chronic inflammatory bowel disease or percutaneous endoscopic gastrostomy
* Patients with stroke mimics:
* Major surgery within the last four weeks
* Myocardial infarction, ischemic stroke, transient ischemic attacks, traumatic brain injury, cerebral venous sinus thrombosis, any intracranial hemorrhage, thrombosis, or pulmonary embolism within the last four weeks
* Chronic inflammatory bowel disease or percutaneous endoscopic gastrostomy
* Healthy subjects:
* Major surgery within the last four weeks
* Myocardial infarction, ischemic stroke, transient ischemic attacks, traumatic brain injury, cerebral venous sinus thrombosis, any intracranial hemorrhage, thrombosis, or pulmonary embolism within the last four weeks
* Chronic inflammatory bowel disease or percutaneous endoscopic gastrostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted with stroke-like symptoms as well as healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 787 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Prediction of clinical outcome as defined by the modified Rankin Scale (mRS) score | 3 months
  The modified Rankin Scale (mRS) is a valid and reliable clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It is a scale used to measure functional recovery (the degree of disability or dependence in daily activities) of people who have suffered a stroke. mRS scores range from 0 (best outcome) to 6 (worst outcome), with 0 indicating no residual symptoms; 5 indicating bedbound, requiring constant care; and 6 indicating death. We will assess associations of clinical outcome with:
  * Global, class, pathway, and individual metabolite levels upon admission (day 1), day 2, day 3, day7, and day 90 [raw values, referenced to HC, or referenced to SM]
  * Global, pathway, and individual protein levels upon admission (day 1), day 2, day 3, day7, and day 90 [raw values, referenced to HC, or referenced to SM]
Prediction of clinical outcome as defined by the modified Rankin Scale (mRS) score | 7 days or day of discharge if earlier (on average 5 days)
  The modified Rankin Scale (mRS) is a valid and reliable clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It is a scale used to measure functional recovery (the degree of disability or dependence in daily activities) of people who have suffered a stroke. mRS scores range from 0 (best outcome) to 6 (worst outcome), with 0 indicating no residual symptoms; 5 indicating bedbound, requiring constant care; and 6 indicating death. We will assess associations of clinical outcome with:
  * Global, class, pathway, and individual metabolite levels upon admission (day 1), day 2, day 3, and day 7 [raw values, referenced to HC, or referenced to SM]
  * Global, pathway, and individual protein levels upon admission (day 1), day 2, day 3, and day 7 [raw values, referenced to HC, or referenced to SM]

SECONDARY OUTCOMES:
Acute brain injury as assessed by neuroimaging | day 1
  The extent of acute brain injury (in ml) will be assessed on admission NCCT and CT perfusion scans.
Subacute brain injury as assessed by neuroimaging | day 3 to day 10
  The extent of subacute brain injury will be manually segmented on images from delayed routine CT or MRI scans.
Neck and cerebral vessel morphology | day 1 to day 10
  We will assess the number of different plaque types on routine CT/MRI angiography scans.
Heart morphology and function as assessed by echocardiography and ECG | day 1 to day 10
  We will assess the likelihood of cardiac embolism by a score that integrates PTFV1, left ventricular strain and left atrial area.
Stroke etiology | 7 days or day of discharge if earlier (on average 5 days)
  Stroke etiology will be assessed using the TOAST classification systems.
Sensitivity and specificity to separet diagnostic groups | day 1 to day 10
  Groups (Ischemic stroke, hemorrhagic stroke, stroke mimics, healthy subjects) will be compared.
Systemic sequelae of stroke | day 1 to day 10
  Systemic sequelae will be assessed by clinical laboratory tests.
Treatment efficacy of mechanical thrombectomy | day 1 to day 90
  Treatment efficacy will be assessed by comparing mRS scores between treated and non-treated groups.

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data, including data dictionaries, that underlie results in a publication, will be made available.
Supporting Information: Analytic Code
Time Frame: IPD and additional supporting information will become available starting 6 months after publication.
Access Criteria: IPD and additional supporting information will be shared with academic researchers with a reasonable request to the corresponding author of the respective publication.